CLINICAL TRIAL: NCT02635425
Title: Aspiration of Limited Number of Eggs to Prevent Severe OHSS in Suspected Cases
Brief Title: Aspiration of Limited Number of Follicles to Prevent Severe Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Hussieny Salama (Other)
Responsible Party: Sponsor-Investigator, Ahmad Hussieny Salama, Associate professor at ainshams university in cairo, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LFOHSS
Record Dates: First submitted 2015-12-12; First posted 2015-12-18 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 eggs collection (Experimental): Aspiration of 7 eggs only
  Interventions: Procedure: 7 eggs collection
- Full eggs collection (Active Comparator): Aspiration of all eggs
  Interventions: Procedure: Full eggs collection

INTERVENTIONS:
Procedure: 7 eggs collection — vaginal US
  Arms: 7 eggs collection
Procedure: Full eggs collection — vaginal US
  Arms: Full eggs collection

SUMMARY:
The purpose of this study is to evaluate the effect of single ovarian puncture to retrieve 7eggs only in prevention of severe ovarian hyperstimulation syndrome.

DETAILED DESCRIPTION:
Thirty patients will be selected for this study grouped into two groups, each group contains fifteen patients.

Group 1 :study group ( retrieval of 7 eggs only). Group 2 :control group ( retrieval of all eggs). Study is held to compare between the two arms, the proportion of patients who will be prevented from the progression to severe OHSS after this interventional method.

ELIGIBILITY:
Inclusion Criteria:

1. More than 9 days of induction of ovulation.
2. Each ovary contains more than 20 follicles.
3. The majority of follicles are >14mm in diameter.
4. Mild fluid in Douglas pouch.
5. The patient started to complain of considerable lower abdominal pains before the egg collection.

Exclusion Criteria:

1. Recurrent ICSI failure or bad obstetric history.
2. Any medical disorder affecting the fluid shift as: diabetes mellitus, autoimmune diseases, hepatic, renal or cardiac conditions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Salama, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 7 Eggs Collection | Full Eggs Collection
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7 Eggs Collection | Full Eggs Collection | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Severe Ovarian Hyperstimulation Syndrome
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | 7 Eggs Collection | Full Eggs Collection
Number analyzed (Participants) | 15 | 15
participants | 2 | 11

ADVERSE EVENTS:
Arm/Group | 7 Eggs Collection | Full Eggs Collection
Serious Adverse Events (participants affected / at risk) | 2/15 | 7/15
Other Adverse Events (participants affected / at risk) | 0/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7 Eggs Collection (N=15) | Full Eggs Collection (N=15)
respiratory depression (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 7 Eggs Collection (N=15) | Full Eggs Collection (N=15)
oliguria (Renal and urinary disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes